CLINICAL TRIAL: NCT01193608
Title: A Phase 1, Multicenter, Randomized, Double-blind, Placebo-controlled, Adaptive, Multiple Ascending Dose Study Of The Safety, Tolerability And Pharmacokinetics Of Aab-003 (Pf-05236812) In Subjects With Mild To Moderate Alzheimer's Disease
Brief Title: Study Evaluating The Safety Of AAB-003 (PF-05236812) In Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2601001; 3245K1-1000 (Other: Alias Study Number)
Record Dates: First submitted 2010-08-19; First posted 2010-09-02 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
Keywords: Randomized; Safety Study; Adaptive; Double Blind
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 0.5 mg/kg AAB-003 (Experimental)
  Interventions: Drug: AAB-003 (PF-05236812)
- 1 mg/kg AAB-003 (Experimental)
  Interventions: Drug: AAB-003 (PF-05236812)
- 2 mg/kg AAB-003 (Experimental)
  Interventions: Drug: AAB-003 (PF-05236812)
- 4 mg/kg AAB-003 (Experimental)
  Interventions: Drug: AAB-003 (PF-05236812)
- 8 mg/kg AAB-003 (Experimental)
  Interventions: Drug: AAB-003 (PF-05236812)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AAB-003 (PF-05236812) — 0.5 mg/kg AAB-003, IV
  Arms: 0.5 mg/kg AAB-003
Drug: AAB-003 (PF-05236812) — 1 mg/kg AAB-003, IV
  Arms: 1 mg/kg AAB-003
Drug: AAB-003 (PF-05236812) — 2 mg/kg AAB-003, IV
  Arms: 2 mg/kg AAB-003
Drug: AAB-003 (PF-05236812) — 4 mg/kg AAB-003, IV
  Arms: 4 mg/kg AAB-003
Drug: AAB-003 (PF-05236812) — 8 mg/kg AAB-003, IV
  Arms: 8 mg/kg AAB-003
Other: Placebo — Placebo, IV
  Arms: Placebo

SUMMARY:
This is a study to evaluate the safety of multiple doses of AAB-003 (PF-05236812) in patients with mild to moderate Alzheimer's Disease. Patients will receive either AAB-003 (PF-05236812) or placebo. Each patient's participation will last approximately 41 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's Disease with MMSE score of 16-26, and brain MRI consistent with the diagnosis of Alzheimer's Disease
* Concurrent use of cholinesterase inhibitor or memantine allowed, if stable.
* Caregiver will participate and be able to attend clinic visits with patient

Exclusion Criteria:

* Significant neurological disease other than Alzheimer's Disease
* Major psychiatric disorder
* Contraindication to undergo brain MRI (e.g., pacemaker, CSF shunt, or foreign metal objects in the body)
* Women of childbearing potential

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (23):
  - Early Phase Investigational Center, Escondido, California
  - Synergy Clinical Research Center of Escondido, Escondido, California
  - MD Clinical, Hallandale, Florida
  - Franck's Pharmacy, Ocala, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Renstar Medical Research, Ocala, Florida
  - Advanced Imaging of Ocala, Ocala, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Foers Medical Arts Pharmacy, Bethesda, Maryland
  - CBH Health, LLC, Rockville, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - KNI/Southwest Michigan Imaging Center, LLC, Kalamazoo, Michigan
  - Brentwood Behavioral Healthcare, Flowood, Mississippi
  - Marty's Pharmacy, Flowood, Mississippi
  - Precise Research Centers, Flowood, Mississippi
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - DePaul Health Center, St Louis, Missouri
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Pharmacare USA, Edison, New Jersey
  - Central Jersey Radiology, Oakhurst, New Jersey
  - Belmont Center for Comprehensive Treatment, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
- South Korea (6):
  - Seoul National University Bundang Hospital, Department of Neurology, Seongnam-si, Gyeonggi-do
  - Inha University Hospital, Department of Neurology, Incheon
  - Samsung Medical Center, Department of Neurology, Seoul
  - Korea University Anam Hospital, Seoul
  - ASAN Medical Center, Seoul
  - Konkuk University Medical Center, Department of Neurology, Seoul

REFERENCES:
- [Derived] Delnomdedieu M, Duvvuri S, Li DJ, Atassi N, Lu M, Brashear HR, Liu E, Ness S, Kupiec JW. First-In-Human safety and long-term exposure data for AAB-003 (PF-05236812) and biomarkers after intravenous infusions of escalating doses in patients with mild to moderate Alzheimer's disease. Alzheimers Res Ther. 2016 Mar 1;8(1):12. doi: 10.1186/s13195-016-0177-y. PMID 26925577
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2601001&StudyName=Study%20Evaluating%20The%20Safety%20Of%20AAB-003%20%28PF-05236812%29%20In%20Subjects%20With%20Alzheimer%27s%20Disease%20

RESULTS

PARTICIPANT FLOW:
Groups:
- AAB-003 0.5 mg/kg: Participants received AAB-003 0.5 milligram/kilogram (mg/kg) 1-hour intravenous (IV) infusion (infusion of AAB-003 and 20 milliliter (mL) normal saline flush of IV line) once every 13 weeks on Day 1, Week 13 and Week 26 for a total of 3 infusions over the course of study. A final follow-up visit was performed at Week 39, 13 weeks after the last infusion.
- AAB-003 1 mg/kg: Participants received AAB-003 1 mg/kg 1-hour IV infusion (infusion of AAB-003 and 20 mL normal saline flush of IV line) once every 13 weeks on Day 1, Week 13 and Week 26 for a total of 3 infusions over the course of study. A final follow-up visit was performed at Week 39, 13 weeks after the last infusion.
- AAB-003 2 mg/kg: Participants received AAB-003 2 mg/kg 1-hour IV infusion (infusion of AAB-003 and 20 mL normal saline flush of IV line) once every 13 weeks on Day 1, Week 13 and Week 26 for a total of 3 infusions over the course of study. A final follow-up visit was performed at Week 39, 13 weeks after the last infusion.
- AAB-003 4 mg/kg: Participants received AAB-003 4 mg/kg 1-hour IV infusion (infusion of AAB-003 and 20 mL normal saline flush of IV line) once every 13 weeks on Day 1, Week 13 and Week 26 for a total of 3 infusions over the course of study. A final follow-up visit was performed at Week 39, 13 weeks after the last infusion.
- AAB-003 8 mg/kg: Participants received AAB-003 8 mg/kg 1-hour IV infusion (infusion of AAB-003 and 20 mL normal saline flush of IV line) once every 13 weeks on Day 1, Week 13 and Week 26 for a total of 3 infusions over the course of study. A final follow-up visit was performed at Week 39, 13 weeks after the last infusion.
- Placebo: Participants received placebo matched to AAB-003 1-hour IV infusion (infusion of placebo matched to AAB-003 and 20 mL normal saline flush of IV line) once every 13 weeks on Day 1, Week 13 and Week 26 for a total of 3 infusions over the course of study. A final follow-up visit was performed at Week 39, 13 weeks after the last infusion.
Period: Overall Study
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Started | 6 | 6 | 16 | 17 | 24 | 19
Completed | 6 | 4 | 14 | 14 | 19 | 17
Not Completed | 0 | 2 | 2 | 3 | 5 | 2
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 3 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized.
Groups:
- AAB-003 0.5 mg/kg: Participants received AAB-003 0.5 mg/kg by IV infusion on Day 1, Week 13 and Week 26
- AAB-003 1 mg/kg: Participants received AAB-003 1 mg/kg by IV infusion on Day 1, Week 13 and Week 26
- AAB-003 2 mg/kg: Participants received AAB-003 2 mg/kg by IV infusion on Day 1, Week 13 and Week 26
- AAB-003 4 mg/kg: Participants received AAB-003 4 mg/kg by IV infusion on Day 1, Week 13 and Week 26
- AAB-003 8 mg/kg: Participants received AAB-003 8 mg/kg by IV infusion on Day 1, Week 13 and Week 26
- Placebo: Participants received placebo matched to AAB-003 by IV infusion on Day 1, Week 13 and Week 26
- Total: Total of all reporting groups
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (6.4) | 67.2 (7.4) | 70.7 (10.8) | 71.5 (8.8) | 64.5 (7.6) | 71.1 (7.6) | 68.6 (8.8)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 3 | 14 | 9 | 14 | 8 | 52
  Male | 2 | 3 | 2 | 8 | 10 | 11 | 36
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 4 | 3 | 5 | 6 | 12 | 11 | 41
  Black | 2 | 2 | 1 | 0 | 1 | 3 | 9
  Asian | 0 | 1 | 10 | 11 | 11 | 5 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Time Frame: Baseline up to 39 Weeks and at Early Withdrawal
Population: Safety analysis set consisted of all participants who received at least one infusion of study medication (including partial infusions). A TEAE was defined as an untoward medical occurrence reported by the participant or investigator following administration of at least one dose of AAB-003.
Measure: Number; unit: Participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Participants
  Participants with Adverse Events (AEs) | 5 | 3 | 10 | 8 | 16 | 12
  Participants with Serious Adverse Events (SAEs) | 1 | 1 | 1 | 0 | 5 | 0
  Participants Discontinued due to AEs | 0 | 0 | 0 | 0 | 3 | 1

2. Primary Outcome: Number of Participants With Laboratory Abnormalities
Time Frame: Baseline up to 39 Weeks and at Early Withdrawal
Population: Safety analysis set consisted of all participants who received at least one infusion of study medication (including partial infusions). Laboratory test parameters included hematology, coagulation, liver function, renal function, electrolytes, clinical chemistry, and urinalysis (dipstick and microscopy).
Measure: Number; unit: Participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Participants | 3 | 3 | 11 | 10 | 12 | 13

3. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Concern
Description: Criteria for potential clinical concern in vital signs included: supine/sitting pulse rate of less than (<) 40 or more than (>) 120 beats per minute (bpm), and standing pulse rate of <40 or >140 bpm; systolic blood pressure (SBP) of more than or equal to (>=)30 millimeters of mercury (mm Hg) change from baseline in same posture and <90 mm Hg; diastolic blood pressure (DBP) >=20 mm Hg change from baseline in same posture and <50 mm Hg. Only supine vital signs were planned for this study. Unplanned sitting vital signs were collected only in the 8/mg and placebo groups and also reported.
Time Frame: Baseline up to 39 Weeks and at Early Withdrawal
Population: Safety analysis set consisted of all participants who received at least one infusion of study medication (including partial infusions).
Measure: Number; unit: Participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Participants
  Supine SBP <90 mm Hg | 0 | 0 | 1 | 0 | 1 | 0
  Maximum increase in supine SBP >=30 mm Hg | 3 | 0 | 3 | 7 | 2 | 6
  Maximum decrease in supine SBP >=30 mm Hg | 0 | 0 | 5 | 0 | 4 | 8
  Sitting SBP <90 mm Hg | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | 0 | 0
  Supine DBP <50 mm Hg | 0 | 0 | 0 | 0 | 0 | 1
  Maximum increase in supine DBP >=20 mm Hg | 2 | 3 | 4 | 2 | 5 | 8
  Maximum decrease in supine DBP >=20 mm Hg | 1 | 0 | 4 | 1 | 4 | 8
  Sitting DBP <50 mm Hg | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | 0 | 0
  Supine pulse rate <40 or >120 bpm | 0 | 0 | 0 | 0 | 0 | 0
  Sitting pulse rate <40 or >120 bpm | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Physical Examination Findings
Time Frame: Baseline up to 39 Weeks and at Early Withdrawal
Population: Safety analysis set consisted of all participants who received at least one infusion of study medication (including partial infusions). A full physical examination consisted of abdomen, genitourinary, cardiovascular systems, lungs, lymph nodes, mouth, musculoskeletal, general, skin, extremities, head, ears, eyes, nose, throat and thyroid.
Measure: Number; unit: Participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Participants | 2 | 4 | 1 | 5 | 9 | 9

5. Primary Outcome: Number of Participants With Abnormal Neurological Examination Findings
Description: The neurological examination was done to the extent needed to assess the participant for any potential changes in neurological status, as determined by the investigator. The minimum items assessed were level of consciousness, speech, cranial nerves, motor, sensory, coordination, gait, and tendon reflexes.
Time Frame: Screening, Day 1 (Baseline) and Weeks 1,6,13,19,26,32, and 39, and at Early Withdrawal
Population: Safety analysis set consisted of all participants who received at least one infusion of study medication (including partial infusions). n = number of evaluable participants at the corresponding time point.
Measure: Number; unit: Participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Participants
  Day 1 (n=6,6,16,17,24,19) | 1 | 2 | 2 | 3 | 1 | 6
  Week 1 (n=6,6,16,17,24,19) | 1 | 1 | 2 | 3 | 0 | 5
  Week 6 (n=6,6,16,17,24,19) | 1 | 1 | 2 | 3 | 0 | 5
  Week 13 (n=6,6,15,16,22,19) | 1 | 1 | 4 | 3 | 0 | 4
  Week 19 (n=6,5,14,15,21,19) | 1 | 1 | 1 | 4 | 1 | 4
  Week 26 (n=6,5,14,14,18,19) | 2 | 1 | 1 | 2 | 1 | 7
  Week 32 (n=6,5,14,14,19,18) | 1 | 1 | 1 | 2 | 0 | 6
  Week 39 (n=6,4,14,14,19,17) | 1 | 1 | 1 | 4 | 0 | 6

6. Primary Outcome: Maximum Observed Serum Concentration (Cmax) for AAB-003 at Day 1
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4 and 6 hours post start of infusion.
Population: Pharmacokinetic (PK) Analysis Set consisted of all randomized participants who received at least one infusion of study medication and have at least one post-dose PK parameter assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24
microgram per milliliter (mcg/mL) | 13.79 (48) | 32.05 (33) | 58.74 (21) | 122.4 (14) | 223.7 (28)

7. Primary Outcome: Maximum Observed Serum Concentration (Cmax) for AAB-003 at at Week 26
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4, 6, and 24 hours post start of infusion.
Population: Evaluable participants in the PK analysis set (all randomized participants who received at least one infusion of study medication and have at least one post-dose PK parameter assessment).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 6 | 5 | 14 | 14 | 17
mcg/mL | 14.53 (33) | 38.51 (25) | 60.17 (38) | 108.5 (41) | 228.9 (30)

8. Primary Outcome: Average Concentration (Cavg) for AAB-003 in Serum at Day 1
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4 and 6 hours post start of infusion.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 6 | 5 | 15 | 16 | 22
mcg/mL | 2.465 (30) | 6.545 (33) | 10.83 (16) | 20.37 (20) | 36.78 (24)

9. Primary Outcome: Average Concentration (Cavg) for AAB-003 in Serum at Week 26
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4, 6, and 24 hours post start of infusion.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 6 | 4 | 14 | 14 | 17
mcg/mL | 3.435 (22) | 7.171 (9) | 12.56 (28) | 22.52 (29) | 46.12 (34)

10. Primary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) for AAB-003 at Day 1
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4 and 6 hours post start of infusion.
Population: PK Analysis Set consisted of all randomized participants who received at least one infusion of study medication and have at least one post-dose PK parameter assessment.
Measure: Median (Full Range); unit: Hours (hr)
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24
Hours (hr) | 1.92 (30) [1.50 to 6.05] | 4.00 (33) [2.17 to 6.02] | 1.54 (16) [1.20 to 2.12] | 1.50 (20) [1.00 to 24.0] | 3.02 (24) [1.07 to 6.00]

11. Primary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) for AAB-003 at Week 26
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4, 6, and 24 hours post start of infusion.
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours (hr)
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 6 | 5 | 14 | 14 | 17
Hours (hr) | 1.56 (22) [1.30 to 4.05] | 2.00 (9) [1.25 to 5.95] | 1.64 (28) [1.05 to 6.03] | 2.00 (29) [1.03 to 6.03] | 1.50 (34) [1.07 to 23.9]

12. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for AAB-003 in Serum at Day 1
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4 and 6 hours post start of infusion.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24
mcg*hr/mL | 5397 (30) | 13470 (33) | 22960 (19) | 44000 (20) | 79130 (23)

13. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for AAB-003 in Serum at Day 1
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4 and 6 hours post start of infusion.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 4 | 3 | 14 | 14 | 19
mcg*hr/mL | 5597 (39) | 13060 (18) | 25270 (17) | 46430 (21) | 82140 (23)

14. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for AAB-003 in Serum at Day 1
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4 and 6 hours post start of infusion.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 6 | 5 | 15 | 16 | 22
mcg*hr/mL | 5384 (30) [1.50 to 6.05] | 14300 (33) [2.17 to 6.02] | 23660 (16) [1.20 to 2.12] | 44490 (20) [1.00 to 24.0] | 80320 (24) [1.07 to 6.00]

15. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for AAB-003 in Serum at Week 26
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4, 6, and 24 hours post start of infusion.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 6 | 4 | 14 | 14 | 17
mcg*hr/mL | 7502 (22) [1.30 to 4.05] | 15660 (9) [1.25 to 5.95] | 27440 (28) [1.05 to 6.03] | 49180 (29) [1.03 to 6.03] | 100700 (34) [1.07 to 23.9]

16. Primary Outcome: Systemic Clearance (CL) for AAB-003 in Serum at Day 1
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4 and 6 hours post start of infusion.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/hour/kilogram (mL/hr/kg)
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 4 | 3 | 14 | 14 | 19
milliliter/hour/kilogram (mL/hr/kg) | 0.08934 (39) | 0.07657 (18) | 0.07914 (17) | 0.08615 (21) | 0.09739 (23)

17. Primary Outcome: Systemic Clearance (CL) for AAB-003 in Serum at Week 26
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4, 6, and 24 hours post start of infusion.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 6 | 4 | 14 | 14 | 17
mL/hr/kg | 0.06665 (22) | 0.06385 (9) | 0.07289 (28) | 0.08133 (29) | 0.07943 (34)

18. Primary Outcome: Volume of Distribution at Steady State (Vss) for AAB-003 in Serum at Day 1
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4 and 6 hours post start of infusion.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 4 | 3 | 14 | 14 | 19
mL/kg | 78.44 (38) | 59.74 (37) | 61.67 (21) | 60.44 (26) | 75.12 (27)

19. Primary Outcome: Volume of Distribution at Steady State (Vss) for AAB-003 in Serum at Week 26
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4, 6, and 24 hours post start of infusion.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 5 | 4 | 13 | 11 | 16
mL/kg | 54.66 (18) | 48.27 (9) | 56.90 (37) | 65.11 (23) | 61.24 (46)

20. Primary Outcome: Serum Decay Half-Life (t1/2) for AAB-003 at Day 1
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4 and 6 hours post start of infusion.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 4 | 3 | 14 | 14 | 19
Days | 27.77 (6.9880) | 20.04 (8.9210) | 24.45 (4.8686) | 21.10 (5.2000) | 22.89 (4.5086)

21. Primary Outcome: Serum Decay Half-Life (t1/2) for AAB-003 at Week 26
Time Frame: Pre-dose, 1 hour (end of infusion), 1.5, 2, 4, 6, and 24 hours post start of infusion.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 5 | 4 | 13 | 11 | 16
Days | 23.41 (6.8638) | 22.32 (3.1454) | 22.83 (4.1356) | 22.27 (3.2448) | 22.81 (4.3455)

22. Primary Outcome: Number of Participants With Categorical Scores on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS assessed whether the participant experienced the following: completed suicide (1), suicide attempt (2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3)("Yes" on "preparatory acts or behavior"), suicidal ideation (4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7)("Yes" on "Has participant engaged in non-suicidal self-injurious behavior").
Time Frame: Baseline up to Week 39 or Early Withdrawal
Population: Safety Analysis Set included all participants who received at least one infusion of study medication (including partial infusions).
Measure: Number; unit: Participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Participants | 0 | 0 | 1 | 0 | 1 | 2

23. Primary Outcome: Number of Participants With New Occurrence of Brain Magnetic Resonance Imaging (MRI) Finding
Description: Brain MRIs were collected during the course of study to assess for any potential drug-related changes that might have constituted a safety concern for study participants. Findings suggestive of either vasogenic edema (VE) or intracranial hemorrhage represented adverse events of special circumstance and were to be reported immediately.
Time Frame: Baseline up to Week 32.
Population: Safety Analysis Set included all participants who received an infusion of study medication (including partial infusions).
Measure: Number; unit: Participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Participants | 0 | 0 | 0 | 0 | 5 | 0

24. Primary Outcome: Number of Participants With Vasogenic Edema of All Severity After Each Infusion Visit
Description: VE of the brain, identified via MRI, was identified as an adverse event of special circumstance.
Time Frame: Day 1, Week 13, and Week 26
Population: Safety Analysis Set included all participants who received an infusion of study medication, including partial infusions. n = number of evaluable participants at the corresponding timeframe.
Measure: Number; unit: Participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Participants
  Day 1 (n=6,6,16,17,24,19) | 0 | 0 | 0 | 0 | 1 | 0
  Week 13 (n=6,5,15,16,21,17) | 0 | 0 | 0 | 0 | 1 | 0
  Week 26 (n=6,5,14,14,17,16) | 0 | 0 | 0 | 0 | 0 | 0

25. Primary Outcome: Number of Participants With Change From Baseline and Absolute Values in Electrocardiogram (ECG) Meeting Categorical Summarization Criteria
Description: Criteria for ECG values of potential clinical concern are: interval between the start of the ECG P wave and the start of the QRS complex corresponding to the time between onset of atrial depolarization and onset of ventricular depolarization (PR): >= 300 milliseconds (msec), and >=25% increase when baseline >=200 msec/ >=50% increase when baseline less than or equal to (<=) 200 msec; time from ECG Q wave to the end of S wave corresponding to ventricular depolarization (QRS): >=200 msec, and >=25% increase when baseline >100 msec/ >=50% increase when baseline <=100 msec; QTc using Fridericia's formula (QTcF) interval: 450 to <480 msec, >=480 msec; QTcF change from baseline: 30 to <60 msec, and >=60 msec.
Time Frame: Baseline, Weeks 1,13,16,26,39 or Early Withdrawal
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Participants
  Maximum PR Interval >=300 msec | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QRS Complex >=200 msec | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QTcF Interval 450 to <480 msec | 0 | 2 | 5 | 4 | 4 | 3
  Maximum QTcF Interval 480 to <500 msec | 0 | 0 | 1 | 0 | 1 | 0
  Maximum QTcF Interval >=500 msec | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval >=25/50% increase | 0 | 0 | 0 | 0 | 0 | 0
  QRS Complex >=25/50% increase | 0 | 0 | 0 | 0 | 0 | 1
  Maximum QTcF Increase from Baseline 30 to <60 msec | 2 | 1 | 2 | 1 | 2 | 3
  Maximum QTcF Interval Increase >=60 msec | 0 | 0 | 0 | 0 | 0 | 0

26. Other Pre Specified Outcome: Number of Participants With Positive Anti-product Antibody Response to AAB-003 in Serum
Description: Human serum anti-drug antibodies (ADA) samples were analyzed for the presence or absence of anti-AAB-003 antibodies by enzyme-linked immunosorbent assay (ELISA) method
Time Frame: Day 1 (predose), Week 13 (predose), Week 26 (predose) and Week 39 or Early Withdrawal
Population: All participants who received an infusion of study medication. n = number of evaluable participants at the corresponding timeframe.
Measure: Number; unit: Participants
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Participants
  Day 1 (n=6,6,16,17,24,19) | 0 | 0 | 0 | 0 | 0 | 0
  Week 13 (n=6,5,15,16,22,19) | 0 | 0 | 0 | 0 | 0 | 0
  Week 26 (n=6,5,14,14,17,18) | 0 | 0 | 0 | 0 | 0 | 0
  Week 39 (n=6,4,14,14,19,16) | 0 | 0 | 0 | 0 | 0 | 0

27. Other Pre Specified Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog) Score at Weeks 13, 26 and 39
Description: The ADAS-cog 70 Point is a structured scale (approximately 40 min to complete) that evaluates memory, orientation, attention, reasoning, language and constructional praxis. This study used the 11-item cognitive subscale of the ADAS-Cog with scores ranging from 0 to 70 points; higher scores indicated greater cognitive impairment.
Time Frame: Baseline, Weeks 13, 26 and 39
Population: All participants who were randomized to a treatment and received at least one infusion of study medication. n = number of evaluable participants at the corresponding timeframe.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Units on a scale
  Baseline (n=6,6,16,17,24,19) | 12.6 (3.73) | 20.4 (7.49) | 21.6 (10.76) | 23.0 (11.15) | 18.0 (7.28) | 18.4 (7.54)
  Week 13 (n=6,5,15,15,22,19) | 1.3 (1.45) | 3.3 (4.39) | -0.4 (5.08) | 3.2 (4.18) | -1.2 (4.20) | 0.2 (3.40)
  Week 26 (n=6,5,14,13,18,19) | 0.9 (2.73) | 0.7 (4.73) | 0.5 (5.40) | 3.3 (5.55) | -0.8 (5.07) | 1.4 (5.85)
  Week 39 (n=6,4,14,13,19,17) | 0.2 (3.13) | 1.4 (3.41) | 2.6 (6.80) | 4.1 (9.80) | -0.5 (5.88) | 1.4 (3.95)

28. Other Pre Specified Outcome: Change From Baseline in Disability Assessment in Dementia (DAD) Score at Weeks 13, 26 and 39
Description: The DAD is a functional assessment based on an interview with the caregiver that takes approximately 20 min to administer and it is comprised of 40 items, 17 related to self-care and 23 items involving instrumental activities of daily living. The DAD is scored from 0 to 100 (higher scores indicate better functioning).
Time Frame: Baseline, Weeks 13, 26 and 39
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Units on a scale
  Baseline (n=6,6,16,17,24,19) | 84.5 (11.27) | 63.7 (31.89) | 78.6 (20.84) | 77.9 (17.91) | 84.8 (15.31) | 84.9 (12.65)
  Week 13 (n=6,6,15,16,22,19) | 5.7 (8.82) | -1.2 (14.22) | -3.8 (11.61) | -5.1 (15.57) | -6.3 (12.71) | -3.0 (7.56)
  Week 26 (n=6,5,14,14,18,19) | 4.3 (9.20) | -0.8 (12.30) | -3.8 (10.20) | -10.4 (14.93) | 0.2 (14.32) | -2.5 (7.73)
  Week 39 (n=6,4,14,14,19,17) | -1.8 (8.40) | 0.5 (12.92) | -6.9 (11.33) | -14.6 (19.52) | -1.9 (12.39) | -1.8 (11.31)

29. Other Pre Specified Outcome: Change From Baseline in Behavioral Symtoms as Measured by the Neuropsychiatric Inventory (NPI) at Weeks 13, 26 and 39
Description: The NPI is an instrument used to assess changes of behavior that have appeared in a defined period of time in participants with Alzheimer's disease (AD) and other dementias. Twelve (12) behavioral areas are assessed in the NPI - delusions, apathy, hallucinations, disinhibition, agitation, irritability, depression, aberrant motor behavior, anxiety, nighttime behaviors, euphoria, appetite, and eating changes. The NPI score is based on frequency and severity of specific behaviors within these categories as reported by the caregiver. A separate caregiver distress score may also be included. The NPI ranges from 0 to 144 (higher scores indicate greater psychopathology).
Time Frame: Baseline, Weeks 13, 26 and 39
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Units on a scale
  Baseline (n=6,6,16,17,23,19) | 11.7 (9.67) | 6.3 (9.18) | 9.1 (8.69) | 10.8 (11.46) | 7.7 (7.30) | 13.8 (12.93)
  Week 13 (n=6,6,15,15,21,18) | -2.7 (4.80) | 4.8 (6.68) | -0.7 (4.27) | 0.4 (7.31) | 0.3 (4.94) | -2.1 (6.81)
  Week 26 (n=6,5,14,14,18,19) | -1.7 (5.24) | 4.8 (4.09) | -1.2 (2.94) | 4.6 (12.17) | 0.3 (6.01) | -3.4 (8.65)
  Week 39 (n=6,3,14,13,19,17) | 0.5 (5.21) | 3.3 (2.52) | 0.6 (6.61) | 4.8 (17.07) | 0.1 (6.70) | -2.6 (10.63)

30. Other Pre Specified Outcome: Change From Baseline on the Clinical Dementia Rating (CDR) Sum of Boxes (CDR-SB) and Global CDR Rating at Weeks 26 and 39
Description: The CDR scale is a clinician-rated dementia staging instrument that tracks the progression of cognitive impairment in the following 6 categories - memory, orientation, judgment and problem solving, involvement in community affairs, home and hobbies, and personal care based on the CDR interview. The CDR is based on discussions between the clinician with the participant and caregiver using a structured format. A global CDR score is established by clinical scoring rules with values of 0 (no dementia), 0.5 (questionable dementia), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia). A more quantitative version of the CDR scale is obtained by summing up the ratings in each of the 6 categories to provide the (CDR-SB). The CDR-SB scale ranges from 0 to 18 where higher score indicates severe dementia.
Time Frame: Baseline, Weeks 26 and 39
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Units on a scale
  CDS-SB - Baseline (n=6,6,16,17,24,19) | 8.00 (1.673) | 11.17 (4.070) | 9.50 (4.351) | 10.94 (3.614) | 8.75 (3.566) | 8.89 (3.381)
  Global CDR - Baseline (n=6,6,16,17,24,19) | 0.67 (0.258) | 1.08 (0.492) | 1.03 (0.618) | 1.09 (0.476) | 0.85 (0.429) | 0.87 (0.467)
  CDR-SB - Week 26 (n=6,5,14,14,18,19) | 1.33 (1.751) | 1.40 (1.517) | -0.07 (2.056) | 1.29 (2.758) | 0.17 (1.855) | 0.16 (1.979)
  Global CDR - Week 26 (n=6,5,14,14,18,19) | 0.33 (0.408) | 0.30 (0.447) | 0.04 (0.414) | 0.25 (0.510) | 0.03 (0.320) | -0.03 (0.262)
  CDR-SB - Week 39 (n=6,4,14,14,19,17) | 1.00 (3.286) | 1.75 (1.708) | 1.00 (2.449) | 1.86 (3.371) | 0.79 (2.840) | -0.35 (1.935)
  Global CDR - Week 39 (n=6,4,14,14,19,17) | 0.33 (0.408) | 0.13 (0.250) | 0.04 (0.414) | 0.50 (0.679) | 0.13 (0.436) | -0.06 (0.300)

31. Other Pre Specified Outcome: Change From Baseline on the Mini Mental State Exam (MMSE) Score at Weeks 13, 26, and 39
Description: The MMSE is a brief 30-point questionnaire test that is used to assess cognition. It is commonly used to screen for dementia. In the time span of about 10 min, it samples various functions, including arithmetic, memory and orientation. Scores range from 0 to 30 (higher scores indicate less impairment) and participants with scores of 16 to 26 were eligible.
Time Frame: Baseline, Weeks 13, 26 and 39
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
Units on a scale
  Baseline (n=6,6,16,17,24,19) | 22.7 (1.37) | 22.5 (2.43) | 20.8 (3.71) | 20.1 (3.00) | 21.2 (2.82) | 21.2 (3.78)
  Week 13 (n=6,6,15,16,22,19) | 1.8 (2.32) | -0.5 (2.35) | 0.1 (2.45) | -1.4 (2.78) | 0.9 (2.00) | 1.0 (1.60)
  Week 26 (n=6,5,14,14,18,19) | 1.8 (1.72) | 0.2 (1.10) | 0.0 (3.51) | -2.0 (2.96) | 1.6 (2.91) | 0.7 (2.91)
  Week 39 (n=6,4,14,14,19,17) | 1.5 (4.18) | -1.0 (0.82) | -0.2 (2.58) | -2.2 (4.56) | 1.4 (3.55) | 0.5 (3.06)

32. Other Pre Specified Outcome: Cerebrospinal Fluid (CSF) Concentration of AAB-003 at Week 32
Description: Participants enrolled in the 2, 4 and 8 mg/kg cohorts participated in an optional CSF collection. Participants enrolled in the maximum tolerated dose (MTD) cohort were mandatorily collected for CSF.
Time Frame: Week 32 or Early Withdrawal
Population: All randomized and treated participants in the 2, 4 and 8 mg/kg cohorts who consented to the collection of CSF samples.
Measure: Mean (Standard Deviation); unit: nanogram/millliter (ng/mL)
Arm/Group | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg
Number analyzed (Participants) | 1 | 1 | 15
nanogram/millliter (ng/mL) | 15.220 (NA) — Standard deviation was not estimable since only one participant was evaluable | 45.020 (NA) — Standard deviation was not estimable since only one participant was evaluable | 79.160 (53.0486)

33. Other Pre Specified Outcome: Change From Baseline in CSF Amyloid-beta x-40 Concentration at Week 32 for AAB-003 8 mg/kg and Placebo Groups
Time Frame: Baseline and Week 32
Population: The CSF analysis set consisted of participants in the AAB-003 8 mg/kg cohort who had provided sufficient CSF samples at Baseline and Week 32 to allow for assaying of both samples, and who had no occurrence of VE.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 15 | 5
picogram/milliliter (pg/mL) | 113.53 (817.270) | 348.64 (1321.047)
Statistical Analysis 1: Comparison: AAB-003 8 mg/kg; Change from baseline, within group; Test type: Superiority or Other; p = 0.599, t-test, 2 sided; Mean change = 113.53, 80% CI 2-sided [-170.30 to 397.35] — One sample paired t-test

34. Other Pre Specified Outcome: CSF Amyloid-beta x-40 Concentration at Baseline and Week 32 for AAB-003 2 mg/kg and 4 mg/kg Groups
Time Frame: Baseline and Week 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | AAB-003 2 mg/kg | AAB-003 4 mg/kg
Number analyzed (Participants) | 1 | 1
picogram/milliliter (pg/mL)
  Baseline | 5685.4 (NA) — There were insufficient numbers of participants for group analysis. | 7413.6 (NA) — There were insufficient numbers of participants for group analysis.
  Week 32 | 5836.1 (NA) — There were insufficient numbers of participants for group analysis. | 8883.2 (NA) — There were insufficient numbers of participants for group analysis.

35. Other Pre Specified Outcome: Change From Baseline in CSF Amyloid-beta x-42 Concentration at Week 32 for AAB-003 8 mg/kg and Placebo Groups
Time Frame: Baseline and Week 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 15 | 5
pg/mL | 48.85 (174.589) | 24.04 (173.610)
Statistical Analysis 1: Comparison: AAB-003 8 mg/kg; Change from baseline, within group; Test type: Superiority or Other; p = 0.297, t-test, 2 sided; Mean change = 48.85, 80% CI 2-sided [-11.79 to 109.48] — One sample paired t-test

36. Other Pre Specified Outcome: CSF Amyloid-beta x-42 Concentration at Baseline and Week 32 for AAB-003 2 mg/kg and 4 mg/kg Groups
Time Frame: Baseline and Week 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AAB-003 2 mg/kg | AAB-003 4 mg/kg
Number analyzed (Participants) | 1 | 1
pg/mL
  Baseline | 485.6 (NA) — There were insufficient numbers of participants for group analysis. | 217.2 (NA) — There were insufficient numbers of participants for group analysis.
  Week 32 | 343.3 (NA) — There were insufficient numbers of participants for group analysis. | 331 (NA) — There were insufficient numbers of participants for group analysis.

37. Other Pre Specified Outcome: Change From Baseline in CSF Tau Concentration at Week 32 for AAB-003 8 mg/kg and Placebo Groups
Time Frame: Baseline and Week 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 15 | 5
pg/mL | -15.26 (110.229) | 67.94 (63.514)
Statistical Analysis 1: Comparison: AAB-003 8 mg/kg; Change from baseline, within group; Test type: Superiority or Other; p = 0.600, t-test, 2 sided; Mean change = -15.26, 80% CI 2-sided [-53.54 to 23.02] — One sample paired t-test

38. Other Pre Specified Outcome: CSF Tau Concentration at Baseline and Week 32 for AAB-003 2 mg/kg and 4 mg/kg Groups
Time Frame: Baseline and Week 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AAB-003 2 mg/kg | AAB-003 4 mg/kg
Number analyzed (Participants) | 1 | 1
pg/mL
  Baseline | 659.6 (NA) — There were insufficient numbers of participants for group analysis. | 856.1 (NA) — There were insufficient numbers of participants for group analysis.
  Week 32 | 739.4 (NA) — There were insufficient numbers of participants for group analysis. | 1115.6 (NA) — There were insufficient numbers of participants for group analysis.

39. Other Pre Specified Outcome: Change From Baseline in CSF P-tau Concentration at Week 32 for AAB-003 8 mg/kg and Placebo Groups
Time Frame: Baseline and Week 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 15 | 5
pg/mL | 1.23 (8.986) | 1.92 (7.755)
Statistical Analysis 1: Comparison: AAB-003 8 mg/kg; Change from baseline, within group; Test type: Superiority or Other; p = 0.603, t-test, 2 sided; Mean change = 1.23, 80% CI 2-sided [-1.89 to 4.35] — One sample paired t-test

40. Other Pre Specified Outcome: CSF P-tau Concentration at Baseline and Week 32 for AAB-003 2 mg/kg and 4 mg/kg Groups
Time Frame: Baseline and Week 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AAB-003 2 mg/kg | AAB-003 4 mg/kg
Number analyzed (Participants) | 1 | 1
pg/mL
  Baseline | 89 (NA) — There were insufficient numbers of participants for group analysis. | 122.7 (NA) — There were insufficient numbers of participants for group analysis.
  Week 32 | 100.3 (NA) — There were insufficient numbers of participants for group analysis. | 140.5 (NA) — There were insufficient numbers of participants for group analysis.

41. Other Pre Specified Outcome: Maximum Observed Plasma Concentration (Cmax) for Amyloid-Beta x-40
Time Frame: Weeks 1, 3, 6, 10, 13 (pre-dose, 1 hour [end of infusion]), Week 26 (pre-dose, 1 hour [end of infusion], 1.5, 2, 4, 6, and 24 hours post start of infusion), and Weeks 32 and 39.
Population: All randomized participants who received at least one infusion of study medication and have at least one postdose pharmacodynamic (PD) parameter assessment. n = number of evaluable participants at the corresponding timeframe.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 16 | 17 | 24 | 19
ng/mL
  Week 1 - Week 13 (n=6,5,14,16,22,19) | 3.321 (50) | 6.959 (29) | 8.202 (19) | 11.89 (10) | 18.03 (19) | 0.3511 (25)
  Week 26 - Week 39 (n=5,4,14,14,17,14) | 1.964 (35) | 3.805 (31) | 3.804 (23) | 7.537 (26) | 12.25 (20) | 0.4689 (84)

42. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Amyloid-Beta x-40
Time Frame: as for outcome 41
Population: All randomized participants who received at least one infusion of study medication, had a Baseline PD parameter assessment and at least one post-dose PD parameter assessment. n = number of evaluable participants at the corresponding timeframe.
Measure: Median (Full Range); unit: Hours
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 5 | 15 | 16 | 22 | 19
Hours
  Week 1 - Week 13 (n=6,5,14,16,22,19) | 24.2 (50) [22.3 to 149] | 24.0 (29) [24.0 to 169] | 24.0 (19) [24.0 to 170] | 166 (10) [24.0 to 238] | 164 (19) [92.2 to 1050] | 168 (25) [0.000 to 2540]
  Week 26 - Week 39 (n=5,4,14,14,17,14) | 2.03 (35) [2.02 to 596] | 2.00 (31) [2.00 to 2.02] | 983 (23) [2.00 to 1080] | 1010 (26) [958 to 1060] | 1010 (20) [1.98 to 1080] | 1030 (84) [0.000 to 2210]

43. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Amyloid-Beta x-40
Time Frame: Baseline; Day 2 (24 hours post start of infusion); Weeks 1, 6, and 13 (pre-dose, 1 hour [end of infusion]), Week 26 (pre-dose, 1 hour [end of infusion], 1.5, 2, 4, 6, and 24 hours post start of infusion), and Weeks 32 and 39.
Population: All randomized participants who received at least one infusion of study medication, had a Baseline PD parameter assessment, at least one post-dose PD parameter assessment, and who had available data for AUClast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 5 | 14 | 16 | 22 | 19
ng*hr/mL | 2664 (31) [22.3 to 149] | 6041 (47) [24.0 to 169] | 7836 (19) [24.0 to 170] | 12970 (17) [24.0 to 238] | 22910 (25) [92.2 to 1050] | 639.7 (23) [0.000 to 2540]

44. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for Amyloid-Beta x-40
Time Frame: as for outcome 43
Population: All randomized participants who received at least one infusion of study medication, had a Baseline PD parameter assessment, at least one post-dose PD parameter assessment, and who had available data for AUCinf. No participants had available data for AUCinf in AAB-003 8 mg/kg and Placebo Groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 1 | 1 | 9 | 2 | 0 | 0
ng*hr/mL | 2916 (NA) — Standard deviation was not estimable since only one participant was evaluable | 5463 (NA) — Standard deviation was not estimable since only one participant was evaluable | 8965 (19) | 12800 (1) |  |

45. Other Pre Specified Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for Amyloid-Beta x-40
Time Frame: as for outcome 41
Population: All randomized participants who received at least one infusion of study medication, had a Baseline PD parameter assessment, and at least one post-dose PD parameter assessment. n = number of evaluable participants at the corresponding timeframe.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 6 | 5 | 15 | 16 | 22 | 19
ng*hr/mL
  Week 1 - Week 13 (n=6,5,14,16,22,19) | 2647 (31) [22.3 to 149] | 6057 (47) [24.0 to 169] | 7854 (19) [24.0 to 170] | 12940 (17) [24.0 to 238] | 22820 (26) [92.2 to 1050] | 631.6 (23) [0.000 to 2540]
  Week 26 - Week 39 (n=5,4,14,14,17,14) | 2614 (32) [2.02 to 596] | 4929 (37) [2.00 to 2.02] | 6119 (31) [2.00 to 1080] | 11910 (26) [958 to 1060] | 19740 (25) [1.98 to 1080] | 798.8 (55) [0.000 to 2210]

46. Other Pre Specified Outcome: Plasma Decay Half-Life (t1/2) for Amyloid-Beta x-40
Time Frame: as for outcome 43
Population: All randomized participants who received at least one infusion of study medication, had a Baseline PD parameter assessment, at least one post-dose PD parameter assessment, and who had available data for t1/2. No participants had available data for t1/2 in AAB-003 8 mg/kg and Placebo Groups.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Number analyzed (Participants) | 1 | 1 | 9 | 2 | 0 | 0
Day | 26.57 (NA) — Standard deviation was not estimable since only one participant was evaluable | 32.14 (NA) — Standard deviation was not estimable since only one participant was evaluable | 30.71 (3.2303) | 29.41 (5.7374) |  |

ADVERSE EVENTS:
Time Frame: Baseline up to 39 weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | AAB-003 0.5 mg/kg | AAB-003 1 mg/kg | AAB-003 2 mg/kg | AAB-003 4 mg/kg | AAB-003 8 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 1/16 | 0/17 | 5/24 | 0/19
Other Adverse Events (participants affected / at risk) | 5/6 | 3/6 | 10/16 | 8/17 | 10/24 | 12/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AAB-003 0.5 mg/kg (N=6) | AAB-003 1 mg/kg (N=6) | AAB-003 2 mg/kg (N=16) | AAB-003 4 mg/kg (N=17) | AAB-003 8 mg/kg (N=24) | Placebo (N=19)
Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebral Microhaemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vasogenic Cerebral Oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AAB-003 0.5 mg/kg (N=6) | AAB-003 1 mg/kg (N=6) | AAB-003 2 mg/kg (N=16) | AAB-003 4 mg/kg (N=17) | AAB-003 8 mg/kg (N=24) | Placebo (N=19)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear Disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tooth Impacted (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Infusion Site Bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 1 | 1
Tooth Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1
Lymph Node Palpable (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Otoscopy Abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 2 | 3 | 2 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Sinus Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gait Disturbance (General disorders) | 0 | 0 | 1 | 2 | 0 | 1
Infusion Site Erythema (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Infusion Site Haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Infusion Site Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Infusion Site Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood Bilirubin Abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bradykinesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 2 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 2
Depressed Mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival Hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deafness Unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Injection Site Swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lacunar Infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Insomina (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Weight Increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mesenteric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Coordination Abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypersexuality (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Calculus Ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal Cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aortic Calcification (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.